CLINICAL TRIAL: NCT06909396
Title: Stress Response and Hemodynamic Changes Associated With Intrathecal Anesthesia Versus Caudal Epidural Anesthesia in Infants Undergoing Laparoscopic Inguinal Herniorrhaphy: Prospective Randomized Control Study
Brief Title: Stress Response and Hemodynamic Changes Associated With Intrathecal Anesthesia Versus Caudal Epidural Anesthesia in Infants Undergoing Laparoscopic Inguinal Herniorrhaphy
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Tanta University (Other)
Responsible Party: Principal Investigator, Manar Mohammed Ismail, Assistant Lecturer of Anesthesiology, Surgical Intensive Care and Pain Medicine, Faculty of Medicine, Tanta University, Tanta, Egypt., Tanta University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Diagnostic
Other Study IDs: 35680/8/22
Record Dates: First submitted 2025-03-27; First posted 2025-04-03 (Actual); Last update posted 2025-04-03 (Actual); Status verified 2025-03

CONDITIONS: Stress Response; Hemodynamic Changes; Intrathecal Anesthesia; Caudal Epidural Anesthesia; Infants; Laparoscopic Inguinal Herniorrhaphy
MeSH Terms: conditions — Fractures, Stress | interventions — Anesthesia, General

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Control group (Active Comparator): Patients received general anesthesia.
  Interventions: Drug: General anesthesia
- Intrathecal group (Experimental): Patients received intrathecal anesthesia.
  Interventions: Drug: Intrathecal Anesthesia
- Caudal block group (Experimental): Patients received caudal epidural anesthesia.
  Interventions: Drug: Caudal block

INTERVENTIONS:
Drug: General anesthesia — Patients received general anesthesia
  Arms: Control group
Drug: Intrathecal Anesthesia — Patients received intrathecal Anesthesia
  Arms: Intrathecal group
Drug: Caudal block — Patients received caudal epidural anesthesia.
  Arms: Caudal block group

SUMMARY:
The aim of this work was to assess stress response and hemodynamic changes associated with intrathecal anesthesia versus caudal epidural anesthesia in infants undergoing laparoscopic inguinal herniorrhaphy.

DETAILED DESCRIPTION:
Inguinal hernia repair is the most frequent surgical procedure in early childhood. Various regional anesthetic techniques have been employed to provide optimum intraoperative and postoperative pain control after this procedure.

Introduced decades ago, the use of intrathecal (spinal) anesthesia and caudal block in procedures for different types of laparoscopic abdominal surgery is safe and efficient.

Caudal block is now frequently used in intraoperative and postoperative analgesia for pediatric surgery. In infants and children, central neuraxial block is an important modality for acute postoperative analgesia in addition to combined anesthesia, the goals of postoperative analgesia in children are pain eradication, expedient recovery to daily activities, and prevention of progression of acute postsurgical pain to chronic pain or hyperalgesia

ELIGIBILITY:
Inclusion Criteria:

* Age from full term one month to one year.
* Both sexes.
* Patients with clinical criteria of laparoscopic inguinal herniorrhaphy.

Exclusion Criteria:

* Refusal of patients' parents.
* Diseases of the central nervous system.
* Patients with metabolic and coagulation defects.
* Pre-term infant.
* Infection at the site of injection.
* Congenital anomaly in vertebral column.
* Patient treated with corticosteroids.
* Patients with respiratory dysfunction.

Ages: 1 Month to 1 Year | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 120 (Actual)
Dates: Start 2023-06-01 (Actual); Primary Completion 2025-01-20 (Actual); Study Completion 2025-01-20 (Actual)

PRIMARY OUTCOMES:
Serum glucose level | 24 hours postoperatively
  Serum glucose level was recorded pre-operative and just postoperative and 6, 12, and 24h postoperatively.

SECONDARY OUTCOMES:
Serum cortisol level | 24 hours postoperatively
  Serum cortisol level was recorded pre-operative and just postoperative and 6, 12, and 24h postoperatively.
Heart rate | Till the end of surgery (Up to 1 hour)
  Heart rate was recorded at baseline, after induction, then every 15 minutes till the end of surgery.
Mean arterial pressure | Till the end of surgery (Up to 1 hour)
  Mean arterial pressure was recorded at baseline, after induction, then every 15 minutes till the end of surgery.
Intraoperative anesthetic consumption | Intraoperatively
  Intraoperative anesthetic consumption of sevoflurane was recorded.
Total analgesics consumption | 24 hours postoperatively
  Intravenous Tramadol 1 mg/kg is administered intravenously in the event that the Face, Legs, Activity, Cry, Consolability (FLACC) score exceeds 4 within the first 24 hours following surgery.

CONTACTS AND LOCATIONS:
Locations (1):
- Tanta University, Tanta, El-Gharbia, Egypt

IPD SHARING:
Plan to Share IPD: Yes
The data will be available upon a reasonable request from the corresponding author after the end of study for one year.
Supporting Information: Study Protocol
Time Frame: After the end of study for one year.
Access Criteria: The data will be available upon a reasonable request from the corresponding author.